CLINICAL TRIAL: NCT00909987
Title: Phase II, Multicenter, Open-label, Non-randomized Study of Neoadjuvant Chemotherapy With Selective Radiotherapy Use in Patients With Intermediate-Risk Cancer of the Rectum Defined by Magnetic Resonance Imaging
Brief Title: Study of Neoadjuvant CT With Selective Radiotherapy in Patients With Intermediate-Risk Cancer Rectum
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol Multidisciplinario del Cancer Digestivo (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEMCAD-0801
Record Dates: First submitted 2009-03-23; First posted 2009-05-29 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-09

CONDITIONS: Rectum Cancer
Keywords: rectum; intermediate risk cancer rectum; neoadjuvant
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Oxaliplatin; Bevacizumab; Radiotherapy; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): Neoadyuvant chemotherapy with XELOX: Xeloda 1000mg/m2/12h dayly, day one in the afternoon until day 15 in the morning; plus oxaliplatin 130mg/m2 (day 1); and Bevacizumab 7.5 mg/kg (day 1)during 3 cycles (each cycle of 3 weeks).
  Followed by a selective use of chemoradiotherapy with radiotherapy (50.4Gy, 28 sesions of 1.8Gy during 5 weeks) plus Xeloda 825mg/m2/12h dayly.
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Drug: Bevacizumab; Radiation: Radiotherapy; Drug: Capecitabine during all Radiotherapy period; Procedure: Total Mesorectal Excision (TME)

INTERVENTIONS:
Drug: Capecitabine — PO 1000 mg/m2 bid during day 1 to 15 for 3 cycles (every cycle has 3 weeks)
  Other Names: Xeloda
Drug: Oxaliplatin — IV 130 mg/m2 during day 1 for 3 cycles (every cycle has 3 weeks)
Drug: Bevacizumab — IV 7.5 mg/Kg during 30 minutes day 1 during 4 cycles (every cycle has 3 weeks)
  Other Names: Avastin
Radiation: Radiotherapy — Total dose 50.4 Gy administered during 28 days (1.8 Gy/day in 5 weeks).
  Other Names: Neoadjuvant Radiotherapy
Drug: Capecitabine during all Radiotherapy period — 825 mg/m2 bid
  Other Names: Xeloda
Procedure: Total Mesorectal Excision (TME) — 4 weeks from the last chemotherapy dose. In those patients who receive radiation TME wil be performed six weeks after

SUMMARY:
Phase II, Multicenter, Open-label, Non-randomized Study of Neoadjuvant Chemotherapy (CAPECITABINE-OXALIPLATIN + BEVACIZUMAB) with Selective Radiotherapy and Chemotherapy with CAPECITABINE Use in Patients with Intermediate-Risk Cancer of the Rectum Defined by Magnetic Resonance Imaging.

DETAILED DESCRIPTION:
XELOX / Bevacizumab will be administrated for 3 cycles over a 9 week period. XELOX without Bevacizumab will be administrated for an additional cycle over a 4 week period. Patients will undergo re-staging within 3 weeks of their 4th cycle of XELOX. This will include MRI of the pelvis. If the reassessment reveals that there has been no disease progression compared to the pre-treatment evaluation and the patient remains a candidate for an R0 resection, the patient will proceed to definitive rectal cancer surgery within 4 weeks from the last chemotherapy dose. If the surgical oncologist's reassessment reveals that the patient is not a candidate for an R0 resection, the patient will proceed to standard pre-operative radiation with synchronous Capecitabine.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥18 years
* Tumor biopsy with histopathologic confirmation of rectal adenocarcinoma as primary histology
* Patient with measurable disease at the baseline visit
* T3 tumor that meets all the following criteria in high-resolution magnetic resonance imaging (MRI) (3-mm slices) of the pelvis: distal border of tumor more than 5cm form the external edge of the anus and below the sacral promontory (located in the anatomy rectum).
* Candidate for complete surgical resection (R0) with sphincter preservation surgery, prior to the administration of any therapy
* Candidate for systemic therapy with XELOX/BVZ
* ECOG: 0-2
* ANC≥1.5 cells/mm3, Hb>8.0 g/dL, platelets>150,000/mm3 in 2 previous weeks
* Patient who signed the informed consent

Exclusion Criteria:

* Stage T4.
* Distant metastases
* Tumor with an intraperitoneal distal border
* Tumor presenting initially in a low location and judged, prior to any treatment, to require abdominoperineal resection
* Previous chemotherapy for colorectal cancer or incomplete recovery from oncologic surgery or other previous major surgery that, in the opinion of the investigator, precludes the use of a combined modality therapy
* Serum creatinine <1.5 ULN
* Patient who has received previous pelvic radiotherapy
* Patient with an uncontrolled infection
* Presence of a high degree of obstruction (intestinal lumen ≤ 1 cm), unless the patient has undergone protective surgical bypass or an endoscopic stent procedure
* Pt with a history of an arterial thromboembolic event during the previous year.This includes angina (stable or unstable),myocardial infarction (MI),cerebrovascular accident (CVA),or other relevant history in the opinion of the investigator.Note: A patient with a history of thrombotic events, such as deep venous thrombosis, pulmonary embolism, MI or ACV, within the 6 months preceding recruitment may be considered for participation in the clinical trial if they are receiving stable doses of anticoagulant therapy. Similarly, patients being anticoagulated for atrial fibrillation or other conditions can participate if they are receiving a stable dosage of anticoagulant therapy. Clinicians must consider the higher risk of therapy with BVZ among patients with a history of thromboembolic disorders so the decision to allow the patients to participate remains at the discretion of the physician
* Previous treatment with another investigational antitumoral therapy in the 30 days prior to beginning treatment
* History of previous malignancy in the past 5 years, excepting basocellular or squamous cell skin cancer, or properly treated cervix cancer in situ
* Woman with a positive pregnancy test in urine or serum during recruitment, prior to the administration of the study medication, or within 72 hours of beginning to take the study medication, or a woman who is nursing
* WOCBP who does not wish to use or cannot use an effective contraceptive method to avoid pregnancy during the complete study period up to 4 weeks after ending the study.Male subjects also must agree to use an effective method of contraception.Note: WOCBP refers to any woman who has experienced menarche and has not undergone successful surgical sterilization or is not postmenopausal (defined as amenorrhea≥12 consecutive months,or women with hormonal replacement therapy and documented serum levels of follicle stimulating hormone).Even women who are using oral, implanted or injectable contraceptive hormones, mechanical products such as an intrauterine device or barrier methods to prevent pregnancy,or who practice abstinence or have a sterile partner, must be assumed to be WOCBP
* Patient with any other condition or concurrent medical or psychiatric disease who,in opinion of the investigator, is not eligible to enter the study
* Known hypersensitivity to any component of the study drug (XELOX/bevacizumab) or radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-03; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of XELOX/BVZ neoadjuvant therapy with selective radiotherapy use in patients with locally advanced tumors of the rectum, measured in terms of the proportion of responders (PCR + CCR), according to RECIST criteria | Until the end of study

SECONDARY OUTCOMES:
Study treatment,which selectively omits neoadjuvant irradiation,can achieve a R0= 90% | At least 3 years for local recurrence and systemic recurrence
Rate of local and systemic recurrence | At least 3 years for local recurrence and systemic recurrence
Toxicity of treatment | At least 3 years for local recurrence and systemic recurrence
Rate of surgical complications during postoperative | At least 3 years for local recurrence and systemic recurrence
Profile of gene expression before neoadjuvant treatment | At least 3 years for local recurrence and systemic recurrence
Complete Phatologic Response (pCR) | 2012
  Complete pathologic response (pCR)estimated according to the number of subjects that showed yPT0N0 divided by the total number of subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Fernández Martos, Oncologist, Study Chair — Instituto Valenciano de Oncología (IVO); Carles Pericay, Oncologist, Study Director — Complejo Sanitario Parc Taulí; Antonieta Salud, Oncologist, Principal Investigator — Hospital Arnau de Villanova (Lérida); Vicente Alonso, Oncologist, Principal Investigator — Hospital Miguel Servet; María José Safont, Oncologist, Principal Investigator — Hospital General Universitario de Valencia; Ruth Vera, Oncologist, Principal Investigator — Hospital de Navarra; Pilar Escudero, Oncologist, Principal Investigator — Hospital Clínico Universitario Lozano Blesa; Joan Maurel, Oncologist, Principal Investigator — Hospital Clinic i provincial de Barcelona; Jorge Aparicio, Oncologist, Principal Investigator — Hospital La Fe; Jaime Feliú, Oncologist, Principal Investigator — Hospital La Paz; Mengual, Radiotherapy, Principal Investigator — Instituto Valenciano de Oncología (IVO); Moisés Miraflores, Radiotherapy, Principal Investigator — Hospital Arnau de Vilanova (Lérida); Martín Tejedor Gutierrez, Radiotherapy, Principal Investigator — Hospital Miguel Servet; Ana Hernández Machancoses, Radiotherapy, Principal Investigator — Hospital General Universitario de Valencia; Fernando Arias de la Vega, Radiotherapy, Principal Investigator — Hospital de Navarra; Javier Valencia, Radiotherapy, Principal Investigator — Hospital Clínico Universitario Lozano Blesa; Carles Conill, Radiotherapy, Principal Investigator — Hospital Clinic i provincial de Barcelona; Alejandro Tormo Micó, Radiotherapy, Principal Investigator — Hospital La Fe; María Elena Sánchez Santos, Radiotherapy, Principal Investigator — Hospital La Paz; Jorge Campos, Surgeon, Principal Investigator — Instituto Valenciano de Oncología (IVO); Enrique Sierra Grañón, Surgeon, Principal Investigator — Hospital Arnau de Vilanova (Lérida); Andrés Monzón, Surgeon, Principal Investigator — Hospital Miguel Servet; José Vicente Roig, Surgeon, Principal Investigator — Hospital General Universitario de Valencia; Javier Suárez Alecha, Surgeon, Principal Investigator — Hospital de Navarra; Eloy Tejero, Surgeon, Principal Investigator — Hospital Clínico Universitario Lozano Blesa; Antonio Lazy, Surgeon, Principal Investigator — Hospital Clinic i provincial de Barcelona; Rafael Estevan, Surgeon, Study Director — Hospital La Fe; Damián García Olmo, Surgeon, Principal Investigator — Hospital La Paz; Jesús Santos, Radiologist, Principal Investigator — Instituto valenciano de Oncología (IVO); Ana Darnell, Radiologist, Study Director — Complejo Sanitario Parc Taulí; Luís Sarriá, Radiologist, Principal Investigator — Hospital Miguel Servet; Vicente Martínez Sanjuán, Radiologist, Principal Investigator — Hospital General Universitario de Valencia; Javier Jiménez, Radiologist, Principal Investigator — Hospital de Navarra; José Antonio Fernández Gómez, Radiologist, Principal Investigator — Hospital Clínico Universitario Lozano Blesa; Juan Ramón Ayuso, Radiologist, Principal Investigator — Hospital Clinic i provincial de Barcelona; Fernando Mas Estellés, Radiologist, Principal Investigator — Hospital La Fe; Paula Alegría Hidalgo, Radiologist, Principal Investigator — Hospital La Paz; Anna Caltrava, Pathologist, Study Director — Instituto Valenciano de Oncología (IVO); Alex Casalots, Pathologist, Principal Investigator — Complejo Sanitario de Parc Taulí; Xavier Matias-Guiu Guia, Pathologist, Principal Investigator — Hospital Arnau de Vilanova (Lérida); Carlos Hörndler, Pathologist, Principal Investigator — Hospital Miguel Servet; Encarna Martínez, Pathologist, Principal Investigator — Hospital General Universitario de Valencia; María Luisa Gómez Dorronsoro, Pathologist, Principal Investigator — Hospital de Navarra; Javier Ortego, Pathologist, Principal Investigator — Hospital Clinico Universitario Lozano Blesa; María José Artes, Pathologist, Principal Investigator — Hospital La Fe; Marta Martín Richard, Oncologist, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Manuel Gallén, Oncologist, Principal Investigator — Hospital del Mar; Javier Gallego, Oncologist, Principal Investigator — Hospital General Universitario de Elche
Locations (12):
- Spain (12):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Barcelona
  - Complejo Sanitario Parc Taulí, Sabadell, Barcelona
  - Hospital Arnau de Vilanova, Lleida, Lérida
  - Hospital La Paz, Madrid, Madrid
  - Hospital de Navarra, Pamplona, Pamplona
  - Hospital La Fe, Valencia, Valencia
  - Instituto Valenciano de Oncología (IVO), Valencia, Valencia
  - Hospital General de Valencia, Valencia, Valencia
  - Hospital Miguel Servet, Zaragoza, Zaragoza

REFERENCES:
- [Derived] Fernandez-Martos C, Brown G, Estevan R, Salud A, Montagut C, Maurel J, Safont MJ, Aparicio J, Feliu J, Vera R, Alonso V, Gallego J, Martin M, Pera M, Sierra E, Serra J, Delgado S, Roig JV, Santos J, Pericay C. Preoperative chemotherapy in patients with intermediate-risk rectal adenocarcinoma selected by high-resolution magnetic resonance imaging: the GEMCAD 0801 Phase II Multicenter Trial. Oncologist. 2014 Oct;19(10):1042-3. doi: 10.1634/theoncologist.2014-0233. Epub 2014 Sep 10. PMID 25209376